CLINICAL TRIAL: NCT00945711
Title: Characteristics of Persons With an Eating Disorder and Type 1 Diabetes and Psychological Comparisons to Persons With an Eating Disorder and No Diabetes
Brief Title: Characteristics of Persons With an Eating Disorder and Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: Park Nicollet Eating Disorder Institute (Other); International Diabetes Center at Park Nicollet (Other); Park Nicollet Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 03802-08-C
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2013-08

CONDITIONS: Eating Disorder; Type 1 Diabetes
Keywords: dual diagnosis
MeSH Terms: conditions — Feeding and Eating Disorders; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Eating Disorder Diabetes Mellitus T1 patients
- 2: Eating Disorder only patients

SUMMARY:
The purpose of this study is to analyze a chart audit of patients seen at Park Nicollet Eating Disorder Institute (EDI) to identify and compare general characteristics of eating disorders with type 1 diabetes patients to a matched eating disordered population without type 1 diabetes, also seen at EDI.

DETAILED DESCRIPTION:
The goal of this study is to conduct a chart audit on all patients with type 1 diabetes who have been seen collaboratively by International Diabetes Center (IDC) and Park Nicollet Eating Disorder Institute (EDI) staff from 2005 - 2008 and their matched eating disordered controls.

Research Questions

1. What are the general characteristics of the ED DM T1 population?
2. How are ED DM T1 patients different from the matched eating disordered patients with respect to race, marital status, age of onset, eating behaviors, self-reported highest and lowest weight, exercise frequency and duration, number of hospital admissions, number of emergency room visits, medication needs, and other medical and psychological/psychiatric comorbidities?
3. How are ED DM T1 patients different from the matched eating disordered patients with respect to the affective and cognitive aspects of eating disorders such as self-reported depression symptoms, body image distortion, thoughts and feelings about eating, psychological concerns, readiness to change, self-esteem and anxiety?
4. For ED DM T1 patients, what is the time relationship of the diagnosis of diabetes and an eating disorder?
5. For ED DM T1 patients, what is the relationship of BMI and A1c?

ELIGIBILITY:
Inclusion Criteria:

* patient seen in both Park Nicollet Eating Disorder Institute and International Diabetes Center for type 1 diabetes from 2005 - 2008
* patient seen only in Park Nicollet Eating Disorder Institute from 2005 - 2008

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Park Nicollet Eating Disorder Institute patient and International Diabetes Center type 1 diabetes patients
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
define general characteristics of the diabetes and eating disorder population | 2005 - 2008

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Powers, PhD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States